CLINICAL TRIAL: NCT06992739
Title: A Prospective, Single-arm Phase II Trial of Trilaciclib Administered Prior to Sacituzumab Tirumotecan in Patients With EGFR-mutated, Advanced Non-Small Cell Lung Cancer (NSCLC) Who Have Progressed on Prior EGFR Tyrosine Kinase Inhibitors（PROTECT-2）
Brief Title: Trilaciclib in Patients Receiving Sacituzumab Tirumotecan for EGFR-mutated, Advanced Non-Small Cell Lung Cancer (NSCLC)
Acronym: PROTECT-2
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PROTECT-2
Record Dates: First submitted 2025-05-06; First posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: NSCLC (Advanced Non-small Cell Lung Cancer); EGFR; Myelosuppression
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — trilaciclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Trilaciclib and Sacituzumab Tirumotecan (Experimental): Trilaciclib and Sacituzumab Tirumotecan
  Interventions: Drug: Trilaciclib and Sacituzumab Tirumotecan

INTERVENTIONS:
Drug: Trilaciclib and Sacituzumab Tirumotecan — Trilaciclib: 240 mg/m2 as a 30-min iv. infusion, completed ≤4h prior to sacituzumab tirumotecan.
  Sacituzumab Tirumotecan: 5 mg/kg on days 1 & 15 of a 28 day cycle via intravenous (IV) infusion until progressive disease or discontinuation.

SUMMARY:
This study is a prospective, single arm phase II clinical trial aimed at patients with advanced non-small cell lung cancer resistant to EGFR-TKI. The aim is to evaluate the efficacy and safety of trilaciclib in bone marrow protection before monotherapy with sacituzumab tirumotecan.

Patients with advanced non-small cell lung cancer resistant to EGFR-TKI, after signing informed consent, will be screened for eligible subjects who meet the inclusion criteria. Prior to receiving treatment with sacituzumab tirumotecan, they will be treated with trilaciclib until disease progression or intolerable toxicity occurs.

Record the dynamic changes of whole blood cell count; Hematological toxicity, including febrile neutropenia and associated infections; Transfusion of blood products and supplementation of hematopoietic raw materials. Perform tumor imaging evaluation according to RECIST 1.1. Baseline imaging examination should be conducted within 21 days prior to the first administration, and tumor imaging evaluation shall be conducted every 6 weeks (± 7 days) from the first study drug administration, or the frequency of imaging evaluation may be increased when there are clinical indications. Subjects who terminate the study drug treatment due to intolerable toxicity or other non disease progression reasons continue to receive tumor evaluation follow-up until disease progression, withdrawal from the study, or death (whichever occurs earliest).

After the screening period and one cycle of treatment, subjects may choose to undergo whole-body PET/CT imaging for exploratory analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Age range: 18-75 years old; No gender restrictions;
2. ECOG PS score 0-1;
3. Expected survival time ≥ 3 months;
4. Patients with locally advanced or metastatic EGFR mutant non-small cell lung cancer diagnosed by histological or cytological examination, who have failed third-generation EGFR-TKI treatment and have experienced up to second-line EGFR-TKI treatment failure;

   1. Patients who have only progressed with 1-2 generations of EGFR-TKI treatment need to undergo third-generation EGFR-TKI treatment;
   2. If patients receive third-generation EGFR-TKI during neoadjuvant and/or postoperative adjuvant therapy and progress to metastatic or locally advanced disease more than 6 months after the last dose, they need to receive third-generation EGFR-TKI treatment again before they can participate in this study;
   3. If patients receive third-generation EGFR-TKI during neoadjuvant and/or postoperative adjuvant therapy and progress to metastatic or locally advanced disease within 6 months after the last dose, they can directly participate in this study;
   4. Imaging disease progression was recorded during or after the recent first-line treatment process.
5. There must be at least one measurable lesion that meets the RECIST 1.1 criteria;
6. The main organ functions well and meets the following standards:

   Blood routine examination (without blood transfusion or correction with hematopoietic stimulating factor drugs within 14 days): hemoglobin (Hb) ≥ 90g/L; Absolute neutrophil count (ANC) ≥ 1.5 × 109/L; Platelet count (PLT) ≥ 80 × 109/L; Biochemical examination: alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN (≤ 5 × ULN for patients with liver metastasis); Serum total bilirubin (TBIL) ≤ 1.5 × ULN (Gilbert syndrome subjects, ≤ 3×ULN）； Serum creatinine (Cr) ≤ 1.5 × ULN, or creatinine clearance rate ≥ 60mL/min; Coagulation function: activated partial thromboplastin time (APTT), international normalized ratio (INR), prothrombin time (PT) ≤ 1.5 × ULN;
7. The subject must recover from all toxic reactions (except hair loss) of previous treatment to ≤ level 1 (evaluated based on CTCAE 5.0 criteria);
8. Women: All women with potential fertility must have a negative serum pregnancy test result during the screening period, and must take reliable contraceptive measures from signing the informed consent form until 3 months after the last dose;
9. Participants voluntarily participate in this study, understand and sign the informed consent form.

Exclusion Criteria:

1. History of myeloid leukemia, myelodysplastic syndrome, or accompanying sickle cell disease;
2. Symptomatic CNS metastases and/or leptomeningeal diseases that require immediate radiotherapy or steroid treatment;
3. Have undergone surgery or radiation therapy within 4 weeks prior to the administration of the first dose of the study drug;
4. Clinical symptoms or diseases of the heart that have not been well controlled, such as: (1) NYHA grade 2 or above heart failure; (2) Unstable angina pectoris; (3) Have experienced myocardial infarction within 6 months; (4) Patients with clinically significant supraventricular or ventricular arrhythmias that require treatment or intervention;
5. History of interstitial lung disease, slow progressive dyspnea and dry cough, sarcoidosis, silicosis, idiopathic pulmonary fibrosis, pulmonary allergic pneumonia, or multiple allergic or peripheral arterial diseases (such as claudication, Leo Buerger's disease).
6. Patients who have received hematopoietic stem cell or bone marrow transplantation in the past;
7. Patients who need to receive radiation therapy at the same time;
8. Those who are known to have a history of allergies to the components of this drug regimen;
9. Pregnant or lactating women;
10. The researcher believes that the patient is not suitable to participate in any other circumstances of this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of grade ≥ 3 neutropenia during sacituzumab tirumotecan treatment | Time from date of first dose of trilaciclib and sacituzumab tirumotecan through 30 days following the last dose of trilaciclib and sacituzumab tirumotecan

SECONDARY OUTCOMES:
Incidence rate of grade 3 or 4 thrombocytopenia | Time from date of first dose of trilaciclib and sacituzumab tirumotecan 30 days following the last dose of trilaciclib and sacituzumab tirumotecan
Incidence rate of grade 3 or 4 anemia during sacituzumab tirumotecan treatment | Time from date of first dose of trilaciclib and sacituzumab tirumotecan through 30 days following the last dose of trilaciclib and sacituzumab tirumotecan
Incidence rate of febrile neutropenia | Time from date of first dose of trilaciclib and sacituzumab tirumotecan through 30 days following the last dose of trilaciclib and sacituzumab tirumotecan
Usage rate of symptomatic treatments for myelosuppression | Time from date of first dose of trilaciclib and sacituzumab tirumotecan through 30 days following the last dose of trilaciclib and sacituzumab tirumotecan
  Such as granulocyte colony-stimulating factor (G-CSF) (not for prevention), thrombopoietin (TPO), interleukin-11 (IL-11), erythropoiesis-stimulating agents (ESA), iron supplements, etc
Objective response rate (ORR) | 18 months after the last subject participating in
Disease control rate (DCR) | 18 months after the last subject participating in
Duration of response (DOR) | 18 months after the last subject participating in
Progression-free survival (PFS) | 18 months after the last subject participating in
Overall survival (OS) | From the date of randomization to the date of death for patients who died in the study due to any cause, or to the last contact date known to be alive for those who survived as of the data cutoff date, assessed up to 30 months.
Incidence rate of adverse events | Time from date of first dose of trilaciclib and sacituzumab tirumotecan through 90 days following the last dose of trilaciclib and sacituzumab tirumotecan
Evaluate the relationship between standardized uptake value (SUV) of target lesion at baseline and treatment efficacy of Sacituzumab Tirumotecan. | 18 months after the last subject participating in
  The changes (%) in lesion SUV values before and after treatment with Sacituzumab Tirumotecan.

IPD SHARING:
Plan to Share IPD: No